CLINICAL TRIAL: NCT00277888
Title: Complications of Jugular and Femoral Venous Catheterization in Critically Ill Patients Requiring Hemodialysis: A Randomized Controlled Trial
Brief Title: Comparison of Femoral Versus Jugular Routes for Temporary Hemodialysis in Seriously Ill Patients
Acronym: CATHEDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHRC-Cathedia
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Kidney Failure, Acute; Critical Illness
Keywords: Dialysis; Hemodialysis; Catheterization
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness | interventions — Renal Dialysis

ARMS (2):
- Femoral route (Experimental)
  Interventions: Procedure: Femoral route for hemodialysis
- Jugular route (Experimental)
  Interventions: Procedure: Jugular route for hemodialysis

INTERVENTIONS:
Procedure: Femoral route for hemodialysis
  Arms: Femoral route
Procedure: Jugular route for hemodialysis
  Arms: Jugular route

SUMMARY:
The purpose of this study is to determine whether a jugular route leads to a lower rate of complications as compared with a femoral route for catheterization in patients admitted in several intensive care units in France who develop acute renal failure requiring hemodiafiltration or hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in intensive care unit (ICU)
* Requiring hemodialysis
* Clinicians have the choice between jugular and femoral routes

Exclusion Criteria:

* Chronic renal failure requiring long term dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2004-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Time of insertion without complication

SECONDARY OUTCOMES:
Rates of mechanical complications
Rates of infectious complications including cath-colonization
Quality of hemodialysis by urea extraction ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Parienti, MD, Principal Investigator — University Hospital, Caen
Locations (10):
- France (10):
  - Medical and nephrologic Intensive Care Unit, CHU Amien Sud, Amiens
  - CH Argenteuil, Argenteuil
  - Medical Intensive Care Unit, CHU de Caen, Caen
  - Surgical Intensive Care Unit, Caen
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU Raymond Pointcarré, Garches
  - Hôpital Cochin, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital St Joseph, Paris
  - CH Saint Malo, St-Malo

REFERENCES:
- [Result] Parienti JJ, Thirion M, Megarbane B, Souweine B, Ouchikhe A, Polito A, Forel JM, Marque S, Misset B, Airapetian N, Daurel C, Mira JP, Ramakers M, du Cheyron D, Le Coutour X, Daubin C, Charbonneau P; Members of the Cathedia Study Group. Femoral vs jugular venous catheterization and risk of nosocomial events in adults requiring acute renal replacement therapy: a randomized controlled trial. JAMA. 2008 May 28;299(20):2413-22. doi: 10.1001/jama.299.20.2413. PMID 18505951
- [Result] Parienti JJ, Megarbane B, Fischer MO, Lautrette A, Gazui N, Marin N, Hanouz JL, Ramakers M, Daubin C, Mira JP, Charbonneau P, du Cheyron D; Cathedia Study Group. Catheter dysfunction and dialysis performance according to vascular access among 736 critically ill adults requiring renal replacement therapy: a randomized controlled study. Crit Care Med. 2010 Apr;38(4):1118-25. doi: 10.1097/CCM.0b013e3181d454b3. PMID 20154599
- [Result] Parienti JJ, Dugue AE, Daurel C, Mira JP, Megarbane B, Mermel LA, Daubin C, du Cheyron D; Members of the Cathedia Study Group. Continuous renal replacement therapy may increase the risk of catheter infection. Clin J Am Soc Nephrol. 2010 Aug;5(8):1489-96. doi: 10.2215/CJN.02130310. Epub 2010 Jun 17. PMID 20558562
- [Result] Dugue AE, Levesque SP, Fischer MO, Souweine B, Mira JP, Megarbane B, Daubin C, du Cheyron D, Parienti JJ; Cathedia Study Group. Vascular access sites for acute renal replacement in intensive care units. Clin J Am Soc Nephrol. 2012 Jan;7(1):70-7. doi: 10.2215/CJN.06570711. Epub 2011 Nov 10. PMID 22076877
- [Result] Parienti JJ, Deryckere S, Megarbane B, Valette X, Seguin A, Sauneuf B, Mira JP, Souweine B, Cattoir V, Daubin C, du Cheyron D; Cathedia Study Group. Quasi-experimental study of sodium citrate locks and the risk of acute hemodialysis catheter infection among critically ill patients. Antimicrob Agents Chemother. 2014 Oct;58(10):5666-72. doi: 10.1128/AAC.03079-14. Epub 2014 Jun 30. PMID 24982071
- [Derived] Iachkine J, Buetti N, de Grooth HJ, Briant AR, Mimoz O, Megarbane B, Mira JP, Ruckly S, Souweine B, du Cheyron D, Mermel LA, Timsit JF, Parienti JJ. Development and validation of a multivariable prediction model of central venous catheter-tip colonization in a cohort of five randomized trials. Crit Care. 2022 Jul 7;26(1):205. doi: 10.1186/s13054-022-04078-x. PMID 35799302
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356
- See also: Guidelines for the prevention of intravascular catheter-related infections — http://www.cdc.gov/mmwr/PDF/rr/rr5110.pdf